CLINICAL TRIAL: NCT07003347
Title: A Randomized, Double-Blind, Placebo Controlled Cross- Over Study to Investigate the Efficacy and Safety of SC0023, a Magnesium Salt Oral Spray Device, in Adults With Refractory or Unexplained Chronic Cough
Brief Title: Study to Investigate the Efficacy and Safety of SC0023, in Adults With Refractory or Unexplained Chronic Cough
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kholood Altassan (Other)
Responsible Party: Sponsor-Investigator, Kholood Altassan, Assistant Professor at Department of Family and Community Medicine, King Saud University
Organization: King Saud University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SC-RCC- KSU001
Record Dates: First submitted 2025-05-14; First posted 2025-06-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral spray of MgCl2 (Experimental)
  Interventions: Device: oral spray of MgCl2
- Placebo (Placebo Comparator)
  Interventions: Device: Saline

INTERVENTIONS:
Device: oral spray of MgCl2 — Magnesium Salt Oral Spray Device
  Arms: oral spray of MgCl2
Device: Saline — oral saline aerosol
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled cross-over study to investigate the efficacy and safety of SC0023 (an oral spray of magnesium based alkaline hypertonic divalent salt) in adults with refractory or unexplained chronic cough over 14 days.

Approximately 20 participants being enrolled and randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18-80 years
* Capable of giving signed informed consent
* Diagnosed with RCC (including unexplained chronic cough) for at least 6 months and at least 4 coughs per hour on average during awake hours at Screening.
* Score ≥ 40 mm on cough severity VAS at screening.
* Normal FEV/FVC
* Women of child-bearing potential must use a highly effective contraception method during the study and for at least 14 days after the last dose.

Exclusion Criteria:

* Current smoker/vaper (all forms of smoking and inhaled substances, including, cannabis/tobacco smoke and nicotine vapors) or individuals who have given up smoking within the past 6 months, or those with >20 pack-year smoking history.
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) bronchiectasis, idiopathic pulmonary fibrosis or uncontrolled asthma.
* Respiratory tract infection within 4 weeks before screening.
* History of malignancy in the last 5 years.
* History of alcohol or drug abuse within the last 3 years.
* Opioid use in last 7 days of screening.
* History of a positive serologic test for, hepatitis B virus surface antigen, or hepatitis C virus.
* Previous participation in clinical trial in last 30 days or 6-half lives of test drug activity.
* Use of prohibited medications anti-tussive therapy, gabapentin, pregabalin, baclofen, tricyclics, systemic corticosteroids, ACE inhibitors, beta blockers.
* Use of dietary supplements containing magnesium for the duration of the study.
* History of myocardial infarction or other cardiac disorders.
* History of any clinically significant or psychiatric condition that in the eyes of the Investigator or designee would not be suitable for this study. Or if in the eyes of the Investigator or designee may prove noncompliant to study procedures.
* Spouses or other family members with a chronic cough in household or
* Living and working in an excessively loud workplace (e.g. building site)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24 hour cough frequency | From Baseline to Day 56

SECONDARY OUTCOMES:
Percentage of participants with a reduction from baseline in the 24-hour cough frequency by ≥ 30%, 50% and 70% compared with placebo. Assessed using HYFE digital cough monitor. | From Baseline to Day 56
Change in cough severity using a visual analogue scale (100 mm visual scale) | From Baseline to Day 56
  100 mm is the worst outcome, 0 is the best outcome.
Patient Global Impression of Change (PGIC, 7-point scale) | From Baseline to Day 56
  Maximum score is 7 and 1 is the minimum score. Higher scores indicate improvement, lower score indicate worsening in condition.
Change in pulmonary lung function test (FEV1 and FVC) | From Baseline to Day 56
Newcastle Laryngeal Hypersensitivity Questionnaire (LHQ) | From Baseline to Day 56
  Score range from 14 to 98. Lower score indicate greater severity.
Safety and Tolerability over 14 days of dosing: a. Incidence (% of subjects) of treatment-emergent adverse events (TEAEs) b. Severity (mild, moderate, or severe) of treatment-emergent adverse events (TEAEs) | 14 Days of Dosing

OTHER OUTCOMES:
Change in exhaled breath condensate (EBC) pH (using an EBC monitor) relative to baseline and placebo over 14 days | 14 Days of Dosing
This study will characterize cough counts over the duration of the study and explore the effect of air quality (where adopted) on cough count and the impact of SC0023 on this parameters. | From Baseline to Day 56
This study will characterize cough counts over the duration of the study and explore the effect of air quality (where adopted) on visual analogue scale (100 mm visual scale) and the impact of SC0023 on this parameters. | From Baseline to Day 56
  100 mm is the worst outcome and 0 mm is the best outcome.
This study will characterize cough counts over the duration of the study and explore the effect of air quality (where adopted) on lung function and the impact of SC0023 on this parameters. | From Baseline to Day 56

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No